CLINICAL TRIAL: NCT05499013
Title: Phase 1/2 Study With an Open-label Dose Escalation Phase Followed by a Randomized, Double-blind Phase of SLN124 in Patients With Polycythemia Vera
Brief Title: Study to Assess SLN124 in Patients With Polycythemia Vera
Acronym: SLN
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Silence Therapeutics plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLN124-004; SANRECO (Other: Silence Therapeutics)
Record Dates: First submitted 2022-07-29; First posted 2022-08-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Polycythemia Vera
Keywords: PV
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Intervention Model Description: Phase 1 is an open-label, dose-finding study. Phase 2 is a randomized, double-blind, placebo-controlled study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 open-label SLN124 (Experimental): SLN124 for subcutaneous (s.c.) injection
  Interventions: Drug: SLN124
- Phase 2 Blinded SLN124 (Experimental): SLN124 for subcutaneous (s.c.) injection
  Interventions: Drug: SLN124
- Phase 2 Blinded Placebo (Placebo Comparator): Sodium chloride for s.c. injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLN124 — SLN124 is a double-stranded small interfering ribonucleic acid (siRNA) targeting transmembrane protease, serine 6 (TMPRSS6) messenger ribonucleic acid (mRNA).
  Arms: Phase 1 open-label SLN124; Phase 2 Blinded SLN124
Drug: Placebo — sodium chloride, solution for injection
  Arms: Phase 2 Blinded Placebo

SUMMARY:
This is a Phase 1/2, multicenter study with an open-label dose escalation followed by a randomized placebo controlled and double-blind phase of SLN124 in adult patients with Polycythemia Vera (PV) to assess the safety, tolerability, efficacy, pharmacokinetic (PK), and Pharmacodynamic (PD) response of SLN124.

ELIGIBILITY:
Phase 1 and Phase 2

Inclusion Criteria:

* Male and female patients aged 18 years or older.
* A confirmed diagnosis of PV according to the revised 2016 World Health Organization criteria:
* Suitable phlebotomy history
* Must agree to adhere to appropriate contraception requirements
* Patients who are not receiving cytoreductive therapy must have been discontinued from any prior cytoreductive therapy for at least 24 weeks before dosing and have recovered from any adverse events due to cytoreductive therapy.
* Patients receiving cytoreductive therapy with hydroxyurea, interferon, busulfan or ruxolitinib must have received a stable dose of cytoreductive therapy for at least 12 weeks before dosing and with no planned change in dose.
* Patients must have had a dermatological examination within 28 weeks prior to dosing.
* Must have an Eastern Cooperative Oncology Group score of 0, 1, or 2.

Exclusion Criteria:

Phase 1 and Phase 2

* Drug intolerance:

  1. History of intolerance to oligonucleotides, or GalNAc, or any component of SLN124.
  2. History of intolerance to s.c. injections.
* Clinically significant thrombosis (e.g., deep vein thrombosis or splenic vein thrombosis) within 12 weeks of screening.
* History of major bleeding events and/or a requirement for blood transfusion therapy owing to bleeding in the last 6 months prior to screening.
* Meets the criteria for post-PV myelofibrosis as defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment
* Any investigational drug less than 6 weeks prior to the first dose of study drug or not recovered from effects of prior administration of any investigational agent.
* Any investigational or marketed product using GalNAc targeting less than 48 weeks prior to administration of any investigational agent (excludes patients with PV who participated in Phase 1 of this study).
* Clinically significant co-morbidities
* Biochemical and hematological parameters:

  1. Biochemical evidence of significant liver disease during screening
  2. Phase 1: Hematological parameters at screening as follows: platelets > 1,000,000/µL; or white blood cell (WBC) count > 25,000/µL; or peripheral blasts > 1%.

  b. Phase 2: Hematological parameters at screening as follows: platelets > 1,000,000/µL; or WBC count > 30,000/µL; or peripheral blasts > 1%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of treatment-emergent adverse events (AEs) | Day 239
  Safety and tolerability will be reported separately following open-label dose escalation phase and double-blind phase
Phase 1: Assessment of the number of phlebotomies at intervals | 6 months prior to dosing to Day 239
Phase 2: Proportion of patients who achieve response between week 18 and week 36 (placebo controlled double blind phase) | 18 to 36 weeks

SECONDARY OUTCOMES:
Phase 1: Pharmacokinetic: area under the plasma concentration (AUC) | Day 127
Phase 1: Pharmacokinetic: peak plasma concentration (Cmax) | Day 127
Phase 1: Pharmacodynamic: change in haematocrit | Day 1 to Day 239
Phase 1: Pharmacodynamic: Change in Transferrin saturation (TSAT) | Day 1 to Day 239
Phase 1: Pharmacodynamic: Change in Hepcidin | Day 1 to Day 239
Phase 2: Comparison of the effect of SLN124 vs placebo | Over 36 weeks
  Number of phlebotomies
Phase 2: Comparison of the effect of SLN124 vs placebo | Over 36 weeks
  Proportion of patients who achieve a response
Phase 2: Comparison of the effect of SLN124 vs placebo | Over 36 weeks
  Safety and tolerability
Phase 2: Comparison of the effect of SLN124 vs placebo | Over 36 weeks
  Hematology parameters and biomarkers of iron metabolism
Phase 2: In the double-blind extension period and in the OLE period: | Week 37 to Week 181
  Assess long-term safety and tolerability of SLN124
Phase 2: In the double-blind extension period and in the OLE period: | Week 37 to Week 181
  Assess long-term effects of SLN124 on QoL assessments
Phase 2: Assessment of SLN124 Cmax at Day 1 and Day 169 of the trial. | Day 1 and Day 169
Phase 2: Assessment of SLN124 PD | Changes from Week 1 to Week 181
  Hepcidin
Phase 2: Assessment of QoL | Changes from Week 1 to Week 181
  MPN-SAF-TSS
Phase 2: Assessment of QoL | Changes from Week 1 to Week 181
  PGI-C
Phase 2: Pharmacodynamic: Change in haematocrit | Changes from Week 1 to Week 181
Phase 2: Pharmacodynamic: Change in Hepcidin | Changes from Week 1 to Week 181

CONTACTS AND LOCATIONS:
Locations (28):
- United States (5):
  - Research Site, Hammond, Louisiana
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Huntsville, Texas
- Australia (7):
  - Research Site, Benowa
  - Research Site, Hobart
  - Research Site, Kurralta Park
  - Research Site 2, Melbourne
  - Research Site, Melbourne
  - Linear Clinical Research, Nedlands
  - Research Site, Richmond
- Bulgaria (2):
  - Research Site 2, Plovdiv
  - Research Site, Plovdiv
- Research Site, Toronto, Canada
- Germany (2):
  - Research Site, Freiburg im Breisgau
  - Research Site, Hanover
- Italy (2):
  - Research Site, Alessandria
  - Research Site, Meldola
- Malaysia (4):
  - Research Site, Johor Bahru
  - Research Site, Kuala Terengganu
  - Research Site, Kuantan
  - Research Site, Kuching
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Lublin
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid